CLINICAL TRIAL: NCT06063512
Title: The Efficacy of Sweet Orange Oil Inhalation in Management of Dental Anxiety and Pain in Children Undergoing Local Anaesthetic Administration: A Randomized Clinical Trial
Brief Title: The Efficacy of Sweet Orange Oil Inhalation in Management of Dental Anxiety and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Abdel Azim Abdel Wahab, Princupal investigator /shaimaa Abdelazim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: aromatherapy in dentistry
Record Dates: First submitted 2023-09-11; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Aromatherapy

STUDY DESIGN:
Intervention Model Description: The two parallel groups will receive the maxillary anaesthesia injection by the same operator.
  In the pre-operative period, MCDAS(f), a self-report measure of anxiety will be recorded for all the children.
  Measuring preoperative dental anxiety (expressed by heart rate) using pulse oximeter
  For Group A (sweet orange oil group): Aromatherapy with inhalers will be carried out, The children will be asked to inhale the aroma from the inhaler For Group B (Control Group): No aromatherapy inhalation . Administration of topical anesthesia . Administration of local anesthesia . After LA administration, Wong-Baker pain rating scale (WBS) will be recorded as a self report measure of pain for all the children.
  After LA administration, anxiety will be recorded again using MCDAS(f) for all the children.
  Measuring postoperative dental anxiety (expressed by heart rate ) using pulse oximeter.
Who Masked: Participant, Investigator
Masking Description: Blinding of the operator and the patients will not be feasible due to the difference between the used techniques. However, the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (sweet orange oil group) (Experimental): Aromatherapy with inhalers will be carried out in an open clinical setting. Three drops of sweet orange oil will be dispensed into a cotton wick of the inhaler, The children will be asked to inhale the aroma from the inhalers for 2 minutes followed by an induction period of 15 minutes.
  Interventions: Other: sweet orange oil inhalation
- For Group B (Control Group) (No Intervention): No aromatherapy inhalation

INTERVENTIONS:
Other: sweet orange oil inhalation — sweet orange oil with inhalers will be carried out in an open clinical setting. Three drops of sweet orange oil will be dispensed into a cotton wick of the inhaler, The children will be asked to inhale the aroma from the inhalers for 2 minutes followed by an induction period of 15 minutes
  Arms: Group A (sweet orange oil group)

SUMMARY:
Aim of the study To evaluate the effectiveness of sweet orange oil inhalation in reducing dental anxiety and pain in children undergoing local anaesthetic administration.

DETAILED DESCRIPTION:
Research Question:

Can sweet orange oil help to overcome dental anxiety and pain in children undergoing local anaesthetic administration?

PICO approach:

* P: Children 8 to 12 years old need dental treatment under local anesthesia.
* I: Sweet Orange oil inhalation.
* C: Without aromatherapy.
* O:

Primary Outcome Dental Anxiety Modified Child Dental Anxiety Scale - Faces version [MCDAS(f)-simplified] Pulse rate

Secondary Outcome

Pain Wong-Baker pain rating scale (WBS)

ELIGIBILITY:
Inclusion Criteria:

* • Children classified with rating 3 (positive) or 4 (definitely positive) according to Frankl behaviour rating scale.

  * Children aged 8-12 years.
  * Patients who need maxillary infiltration anaesthesia in the first dental visit.

Exclusion Criteria:

* Children with any neurological or psychological disorders.

  * Children with previous LA administration.
  * Presence of dental or medical emergency.
  * Presence of systemic disorders.
  * Chidren with common cold.
  * Children with known allergy to topical or local anesthetic agents.
  * Parental refusal for participation.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Through study completion , within 10 months
  Pulse rate
Anxiety | Through study completion , within 10 months
  Modified child dental anxiety scale

SECONDARY OUTCOMES:
Dental pain | Through study completion , within 10 months
  Wong Baker pain rating scale

REFERENCES:
- [Background] Nirmala K, Kamatham R. Effect of Aromatherapy on Dental Anxiety and Pain in Children Undergoing Local Anesthetic Administrations: A Randomized Clinical Trial. J Caring Sci. 2021 Aug 23;10(3):111-120. doi: 10.34172/jcs.2021.026. eCollection 2021 Aug. PMID 34849354